CLINICAL TRIAL: NCT03168165
Title: The Effectiveness of Training Physical Therapists in Pain Neuroscience Education on Patient Reported Outcomes for Patients With Chronic Spinal Pain
Brief Title: PNE Effectiveness Cluster Trial
Acronym: PNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Elizabeth Lane, DPT, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00097154
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Neck Pain; Low Back Pain; Chronic Pain
MeSH Terms: conditions — Neck Pain; Low Back Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care, no intervention
- Pain Neuroscience Education Training (Experimental): The region of clinics randomized to this arm will receive PNE education, which consists of 6 weeks online training followed by an on-site training day.
  Interventions: Other: Pain neuroscience education training

INTERVENTIONS:
Other: Pain neuroscience education training — PNE training will consist of 6 weeks online training followed by one day training session.
  Arms: Pain Neuroscience Education Training

SUMMARY:
This is a cluster randomized trial that involves training regions of physical therapy clinics to use pain neuroscience education or continue with usual care. The investigators will examine outcomes for patients with chronic neck or back pain.

DETAILED DESCRIPTION:
Chronic spinal pain is a very common and costly condition. An estimated 26.4% of Americans have experienced an episode low back pain (LBP) and 13.8% have experienced neck pain in the past 3 months. Lifetime prevalence of spinal pain ranges from 54% to 80% and the estimated healthcare costs for those with spinal pain are 57% higher than those without. While many with acute LBP have a favorable prognosis, those who develop chronic pain continue will experience persistent poor health and place a large burden on the healthcare system.

With growing healthcare costs and mounting disability, there is increased demand for physical therapists to promote more effective self-management strategies for patients with chronic spinal pain. Education is a critical component of self-management. Pain neuroscience education (PNE) is an education method used by physical therapists to help patients understand the biology, physiology and psychological factors influencing their pain experience and to reconcile faulty cognitions and beliefs associated with persistent pain and disability8. PNE has been shown to have positive effects on patient-reported outcomes for a variety of spinal pain conditions. This study will examine the impact of widespread implementation of PNE into routine physical therapy care.

The proposed mechanism of PNE is proposed to relate changes in patients' conceptualization of the pain experience, specifically concepts associated with fear, knowledge, and beliefs of pain. Additional research has identified autonomous motivation and self-efficacy as relevant to patients' behavioral responses to pain. Autonomous motivation is proposed to be an essential factor for behavior change, adhering to a treatment program and persistent positive health behavior changes. Autonomous motivation has not been examined as an influencing factor in the PNE model. Self-efficacy relates to the degree an individual feels they have control over their situation; and high self-efficacy has been associated with more active coping efforts. This study will examine self-efficacy and autonomous motivation as potential mediators of the ability of a PNE intervention improve functional outcomes in a pragmatic clinical environment.

This project's overall goal is to determine the effectiveness of providing physical therapists with PNE training on patient-centered outcomes (physical function and pain interference) for patients with chronic neck or back pain receiving physical therapy. Secondarily, the investigators will explore mechanisms of effects of PNE by examining the role of autonomous motivation and self-efficacy. To accomplish these goals, the investigators will conduct a cluster-randomized clinical trial, randomly assigning groups of clinics to receive PNE training or usual care with no additional training for physical therapists working in the clinic. This design allows for maximum external validity and generalizability across outpatient physical therapy clinics.

Primary Aims I. Compare effectiveness of PNE training vs. no additional training for physical therapists on patient-centered outcomes (physical function and pain interference) for patients with chronic spinal pain. The investigators hypothesize patients receiving treatment from physical therapists receiving PNE education will show greater improvement in patient-centered outcomes.

Secondary Aims I. Compare the effects of PNE training vs. no additional training for physical therapists on the patient-physical therapist alliance. The investigators hypothesize patients receiving treatment from physical therapists receiving PNE education will show greater alliance with their physical therapist.

II. Explore the mediating effects of autonomous motivation and self-efficacy on patient-centered outcomes. The investigators hypothesize autonomous motivation and/or self-efficacy will mediate the effects of education on patient-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 at time of first physical therapy session
* Primary reason for physical therapy is low back and/or neck pain
* Meets the NIH definition of chronic pain (i.e., neck or back pain on at least half the days in the past 6 months.)

Exclusion Criteria:

* No spinal surgery within the previous 12 months
* No evidence of "red flag" conditions (e.g., cauda equine syndrome, cancer, fracture, infection or systemic disease) that requires immediate referral from physical therapy to medical care
* Not currently known to be pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function | 2 week and 12 week
  Change score of Physical Function scores from baseline

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference | 2 week and 12 week
  Change score of Pain Interference scores from baseline
pain self-efficacy | 2 week and 12 week
  Measured by Pain Self-Efficacy Questionnaire
Autonomous motivation | 2 week and 12 week
  Measured by Treatment Self-regulation Questionnaire
Therapeutic Alliance | 2 week and 12 week
  As measured by Working Alliance Theory of Change Inventory

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - BenchMark, Birmingham, Alabama
  - BenchMark, Helena, Alabama
  - BenchMark, Hoover, Alabama
  - BenchMark, Moody, Alabama
  - BenchMark, Phenix City, Alabama
  - Benchmark Physical Therapy, Acworth, Georgia
  - BenchMark, Alpharetta, Georgia
  - BenchMark, Atlanta, Georgia
  - BenchMark, Austell, Georgia
  - BenchMark, Canton, Georgia
  - BenchMark, Carrollton, Georgia
  - BenchMark, Cartersville, Georgia
  - BenchMark, Columbus, Georgia
  - BenchMark, Dallas, Georgia
  - BenchMark, Decatur, Georgia
  - BenchMark, Dunwoody, Georgia
  - BenchMark, Hiram, Georgia
  - BenchMark, Jasper, Georgia
  - BenchMark, Kennesaw, Georgia
  - Rehab South, Lawrenceville, Georgia
  - BenchMark, Marietta, Georgia
  - Rehab South, Newnan, Georgia
  - Rehab South, Peachtree City, Georgia
  - BenchMark, Peachtree City, Georgia
  - BenchMark, Roswell, Georgia
  - BenchMark, Smyrna, Georgia
  - BenchMark, Suwanee, Georgia
  - BenchMark, Tucker, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lane E, Magel JS, Thackeray A, Greene T, Fino NF, Puentedura EJ, Louw A, Maddox D, Fritz JM. Effectiveness of training physical therapists in pain neuroscience education for patients with chronic spine pain: a cluster-randomized trial. Pain. 2022 May 1;163(5):852-860. doi: 10.1097/j.pain.0000000000002436. PMID 34354017
- [Derived] Lane E, Fritz JM, Greene T, Maddox D. The effectiveness of training physical therapists in pain neuroscience education on patient reported outcomes for patients with chronic spinal pain: a study protocol for a cluster randomized controlled trial. BMC Musculoskelet Disord. 2018 Oct 25;19(1):386. doi: 10.1186/s12891-018-2269-2. PMID 30360762